CLINICAL TRIAL: NCT01582087
Title: Evaluation of Mechanisms Responsible for Coma in Patients Affected by Fulminant, Acute and Chronic Hepatic Failure
Status: Terminated | Type: Observational
Why Stopped: At the request of the PI, the Collaborating PI left the university
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Other Study IDs: 12-030
Record Dates: First submitted 2012-04-18; First posted 2012-04-20 (Estimated); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Acute and Chronic Hepatic Failure With Developing Coma
Keywords: acute hepatic failure; chronic hepatic failure; coma
MeSH Terms: conditions — Liver Failure, Acute; End Stage Liver Disease; Coma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Samples previously collected for diagnostic use which could include blood, urine, bile, cerebral spinal fluid, feces, liver tissue, brain tissue.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- acute or chronic hepatic failure: All patients presenting at University of Texas Medical Branch (UTMB) with acute and chronic hepatic failure and who are developing coma

SUMMARY:
The purpose of this study is to understand mechanisms associated with the development of coma during hepatic failure. As of today, those mechanisms are not understood and it is difficult to intervene and prevent coma development which is often associated with mortality. Understanding the mechanism involved, may allow us to prevent coma and develop new therapies to treat this disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients (male or female), 18 years or older hospitalized or seen at UTMB clinics for chronic or acute hepatic failure will be included in the study.

Exclusion Criteria:

* Patients (male or female), 18 years or older hospitalized or seen at UTMB clinics that do not have a diagnosis of chronic or acute hepatic failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: GI clinic hospital inpatient stay
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2018-07-24 (Actual); Study Completion 2018-07-24 (Actual)

PRIMARY OUTCOMES:
The relationship that exist between a liver undergoing chronic or acute degeneration and hepatic coma. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Luca Cicalese, MD, Principal Investigator — The University of Texas Medical Branch
Locations (1):
- The University of Texas Medical Branch, Galveston, Texas, United States